CLINICAL TRIAL: NCT03660163
Title: Assessment of the Outcome of Endodontic Treatment Using Cone Beam Computed Tomography-A Prospective Study
Brief Title: Assessment of the Outcome of Endodontic Treatment Using Cone Beam Computed Tomography.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H0804/79 v.3
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Periapical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the correlation between pre-obturation bacterial detection using fluorescence amplification and outcome of endodontic treatments. Thus, enabling a suitable detection threshold to predict the likelihood of treatment failure. This has the potential to be used a bench side tool in general dental practice to act as a surrogate endpoint for clinicians performing root canal treatment.

DETAILED DESCRIPTION:
Pre-obturation root canal samples were taken using paper points from patients undergoing primary root treatments. The samples were analyzed using a fluorescent spectrometer and a molecular fluorescent vital dye (Calcein AM).

Pre-operative and 1-year post-operative periapical radiographs and Cone Beam Computed Tomography (CBCT) scans were assessed by two calibrated expert examiners to evaluate the outcome of the root canal treatments.

The use of a chairside bacterial stain can allow the clinician to predict the outcome of treatment with confidence. Sampling the root canal space with endodontic paper points followed by ex-situ fluorescent staining and analysis provides a patient-friendly, simple to use and rapid way of predicting root canal treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one tooth diagnosed with the endodontic disease.
* teeth that were tender to percussion and palpation.
* teeth that had a sinus tract and/ swelling.
* Both primary treatment teeth and teeth which had already been root treated were considered.

Exclusion Criteria:

* Patients were excluded if they were pregnant.
* Immunosuppressed patients.
* Non-restorable teeth.
* Teeth with a periodontal probing depth greater than 3mm.
* Teeth with apical radiolucencies with the longest dimension above 1.2cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the endodontic postgraduate unit at Guy's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Periapical periodontium health | One year
  Assess the health of periapical periodontium of a tooth by examining the CBCT image

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Patel, PhD, Principal Investigator — King's College London

REFERENCES:
- [Derived] Knight A, Blewitt I, Al-Nuaimi N, Watson T, Herzog D, Festy F, Patel S, Foschi F, Koller G, Mannocci F. Rapid Chairside Microbial Detection Predicts Endodontic Treatment Outcome. J Clin Med. 2020 Jul 3;9(7):2086. doi: 10.3390/jcm9072086. PMID 32635158